CLINICAL TRIAL: NCT04846621
Title: Comparative Study Between Nicorandil and Nifedipine for the Treatment of Patients Presenting by Preterm Labor
Brief Title: Comparative Study Between Nicorandil and Nifedipine for the Treatment of Preterm Labour
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Ain Shams University (Other)
Responsible Party: Principal Investigator, Manella fayez, Miami, Alexandria Egypt, Ain Shams University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: preterm labor tocolysis
Record Dates: First submitted 2021-04-07; First posted 2021-04-15 (Actual); Last update posted 2021-04-15 (Actual); Status verified 2021-04

CONDITIONS: Preterm Labor With Preterm Delivery
MeSH Terms: interventions — Calcium Channel Blockers

STUDY DESIGN:
Who Masked: Participant
Masking Description: all cases in both groups will not know which drug they receive
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- group Nicorandil (Other): women will receive oral Nicorandil 20 mg initially followed by 10 mg at 8 hourly intervals for 48 hours
  Interventions: Drug: Potassium Channel Opener
- group Nifedipine (Other): Women will receive oral Nifedipine loading dose 20 mg orally followed by 10 mg every 8 hours for 48 hours
  Interventions: Drug: Calcium channel blocker

INTERVENTIONS:
Drug: Potassium Channel Opener — Randomized Controlled comparative clinical trial between two drugs as a tocolytic agent in preterm labor
  Arms: group Nicorandil
Drug: Calcium channel blocker — Randomized Controlled comparative clinical trial between two drugs as a tocolytic agent in preterm labor
  Arms: group Nifedipine

SUMMARY:
Nicorandil (potassium channel activator) is claimed to be as effective as Nifedipine (calcium channel blocker) for tocolysis in preterm labour

aim of the study: To assess the efficacy of Nicorandil compared with Nifedipine as a tocolytic agent in delaying labour for 48 hours following their administration

DETAILED DESCRIPTION:
Preterm labour refers to a delivery that occurs between 20 weeks and before completing 37 weeks of gestation. It may or may not be preceded by preterm labor Preterm labor (PTL) is one of the leading causes of perinatal morbidity and mortality. It is one of the major public health problems, especially with reference to mortality, disability and health care expenses

The diagnosis of preterm labor based upon clinical criteria of regular painful uterine contractions occurs between 20 weeks and before 37 weeks gestation accompanied by cervical change (dilation and/or effacement). Vaginal bleeding and/or ruptured membranes in this setting increase diagnostic certainty , using the following specific criteria:

Uterine contractions (≥4 every 20 minutes or ≥8 in 60 minutes) Plus one of the following:-

* Cervical dilation equal or more than 3 cm
* Cervical length less than 20 mm on transvaginal ultrasound
* Cervical length between 20 to less than 30 mm on transvaginal ultrasound and positive fetal fibronectin test . (This criterion will not be relied upon in this study because it is costly and widely not available in most laboratories)

Since uterine contractions are the most frequently recognized sign of preterm labor, inhibition of uterine contractions with tocolytic agents to prolong pregnancy and reduce neonatal complications has been and continues to be the focus of treatment of preterm labor

• Nifedipine, a calcium channel blocker, could be used as a first line tocolytic agent

Owing to this side effects of Nifedipine, another novel drug (Nicorandil) is studied and according to literature Nicorandil is as effective as Nifedipine for tocolysis in preterm labour

is an anti-angina medication that has the dual properties of a nitrate and ATP-sensitive K+ channel activator. Nicorandil has proved to be safe as anti angina treatement in pergnency

ELIGIBILITY:
Inclusion Criteria:

* BMI between (20 - 30 kg /m²).
* pregnant female with single viable fetus who presented to the outpatient clinic or Emergency room with the criteria of diagnosis of preterm labor between 28 and before completing 34 weeks pregnancy

Exclusion Criteria:

* - Any condition in which continuation of pregnancy will jeopardize maternal or fetal welfare.
* Cervix dilatation greater than 4 cm.
* Polyhydramnios [amniotic fluid index (AFI) greater than 24 cm or deep vertical pocket more than 8 cm.]
* Oligohydramnios (AFI less than 5 cm).
* Suspected intrauterine infection if Maternal fever is present as a constant feature plus one or more of the following:-

  * Maternal leucocytosis (more than 15,000)
  * purulent vaginal discharge
  * Fetal tachycardia more than 180 bpm.
* Growth restriction.
* Major antepartum hemorrhage
* Major maternal medical disorders such as diabetes, hypertension, systemic lupus,liver and kidney dysfunction .
* Multiple gestation pregnancy.
* Signs of fetal non reassuring CTG
* Signs of fetal abnormal CTG
* Lethal fetal anomaly incompatible with life.
* Premature Rupture of membrane.

  --Contraindication for the use of Nifedipine and/or Nicorandil such as drug allergy, cardiac disease, liver disease and kidney disease
* previous caesarean section

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 230 (Estimated)
Dates: Start 2020-06-01 (Actual); Primary Completion 2021-06 (Estimated); Study Completion 2021-07-01 (Estimated)

PRIMARY OUTCOMES:
Number of participants with successful prolongation of pregnancy for a period of 48 hours following administration of the studied drug. | 48 hours prolongation of pregnancy after starting the studied drug
  By follow up of the patients labor progress by the investigator through vaginal examination of the cervical dilatation

SECONDARY OUTCOMES:
assess safety of the drug on fetal outcome | 5 minutes
  By recording the ABGAR score at 1 and 5 minutes after Birth

CONTACTS AND LOCATIONS:
Overall Officials: manella beshara, master, Principal Investigator — Ain Shams University
Locations (1):
- Manella Fayez Zaki Beshara, Egypt, Alexandria Governorate, Egypt

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, ICF
Time Frame: in about 3 months

REFERENCES:
- [Derived] Wilson A, Hodgetts-Morton VA, Marson EJ, Markland AD, Larkai E, Papadopoulou A, Coomarasamy A, Tobias A, Chou D, Oladapo OT, Price MJ, Morris K, Gallos ID. Tocolytics for delaying preterm birth: a network meta-analysis (0924). Cochrane Database Syst Rev. 2022 Aug 10;8(8):CD014978. doi: 10.1002/14651858.CD014978.pub2. PMID 35947046